CLINICAL TRIAL: NCT01803360
Title: A Randomized, Double-blind, Placebo Controlled Trial to Assess the Efficacy of Neridronate 100 mg -4 i.v. Infusions- in Patients With Painful Osteoarthritis of the Knee With Bone Marrow Lesions.
Brief Title: Efficacy Study of Neridronate to Treat Painful Osteoarthritis of the Knee With Bone Marrow Lesions.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Massimo Varenna, MD PhD, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NERI-OA-2013
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — 6-amino-1-hydroxyhexane-1,1-diphosphonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Neridronate (Experimental): Neridronate 100 mg solution for infusion: 4 intravenous administrations in a course of 10 days treatment
  Interventions: Drug: Neridronate
- Placebo (Placebo Comparator): Saline solution for infusion: 4 intravenous administrations in a course of 10 days treatment

INTERVENTIONS:
Drug: Neridronate — Neridronate 100 mg solution for infusion: 4 intravenous administrations in a course of 10 days treatment
  Arms: Neridronate

SUMMARY:
The purpose of this study is to determine whether neridronate is effective in the treatment of pain related to bone marrow oedema in patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of knee Osteoarthritis (ACR criteria)
* Radiographic diagnosis of knee Osteoarthritis (Kellgren/Lawrence scale >=2)
* >4 weeks but <3 months pain, reported as >30 mm on a 100 mm VAS scale
* bone marrow oedema of the affected knee on magnetic resonance

Exclusion Criteria:

* inflammatory arthritis
* aseptic osteonecrosis of the knee
* previous or current treatment with Bisphosphonates
* serum calcium or creatinine abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-07 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
knee pain reduction | 60 days
  to assess the efficacy in terms of proportion of patients with a 50% reduction in pain intensity compared to baseline measured by VAS 100 mm scale recorded at the last visit (day 60)

SECONDARY OUTCOMES:
Bone marrow lesions reduction | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Gaetano Pini, Milan, MI, Italy

REFERENCES:
- [Derived] Varenna M, Zucchi F, Failoni S, Becciolini A, Berruto M. Intravenous neridronate in the treatment of acute painful knee osteoarthritis: a randomized controlled study. Rheumatology (Oxford). 2015 Oct;54(10):1826-32. doi: 10.1093/rheumatology/kev123. Epub 2015 May 20. PMID 25998450